CLINICAL TRIAL: NCT03825588
Title: As Safe As Possible (ASAP): A Balanced, Two-by-Two Design To Test Conjoint and Unique Efficacy of an Inpatient Intervention and an Emotion Regulation/Safety Planning App in Preventing Suicide Attempts Post-Discharge
Brief Title: Establishing Efficacy of an Inpatient Intervention and Phone App to Reduce Suicidal Risk
Acronym: ASAP+BRITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: University of Pittsburgh (Other); American Foundation for Suicide Prevention (Other)
Responsible Party: Principal Investigator, Beth Kennard, PROFESSOR, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: STU 112016-057
Record Dates: First submitted 2018-12-10; First posted 2019-01-31 (Actual); Results first posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Suicidal Ideation; Suicide, Attempted
MeSH Terms: conditions — Suicidal Ideation; Suicide, Attempted | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Investigators will randomize 240 hospitalized suicidal adolescents with a history of a suicide attempt or ideation with plan to one of 4 conditions in a 2 by 2 design: (1) ASAP + BRITE; (2) BRITE + TAU (treatment as usual); (3) ASAP + TAU; or (4) TAU alone to determine the single and additive effects of ASAP and BRITE on suicide attempts in the subsequent six months.
Who Masked: Outcomes Assessor
Masking Description: During the RCT, the independent evaluator (IE) will be blinded to the assigned condition and will take the following steps to preserve the blind: participants and families will be asked not to share with the IE which condition they are assigned to; at staff meetings when cases are reviewed, IEs will not be present; IEs will be asked to guess what the treatment assignment is at the end of each interview, and they will notify the project coordinator if they become unblinded. Participants will complete complementary self-report forms that will not be influenced by interviewer bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ASAP + BRITE + TAU (treatment as usual) (Experimental): Participants in this arm receive the ASAP (As Safe As Possible) intervention, during their transition from inpatient to outpatient care, as well as the BRITE smart phone app for distress tolerance/emotion regulation and safety planning. Participants will also receive usual treatment protocols that all adolescents admitted to their respective Inpatient Psychiatry program receive. Participants complete paper safety plans as part of their regular treatment, which is a standard of care for suicidal youth.
  Interventions: Behavioral: ASAP (As Safe As Possible); Behavioral: BRITE smart phone app; Behavioral: TAU (treatment as usual)
- BRITE + TAU (treatment as usual) (Experimental): Participants in this arm will receive the BRITE smart phone app for distress tolerance/emotion regulation and safety planning as they proceed from inpatient to outpatient care, in addition to usual treatment protocols that all adolescents admitted to their respective Inpatient Psychiatry program receive. Participants complete paper safety plans as part of their regular treatment, which is a standard of care for suicidal youth.
  Interventions: Behavioral: BRITE smart phone app; Behavioral: TAU (treatment as usual)
- ASAP + TAU (treatment as usual) (Experimental): Participants in this arm will receive the ASAP (As Safe As Possible) intervention during their transition from inpatient to outpatient care, in addition to usual treatment protocols that all adolescents admitted to their respective Inpatient Psychiatry program receive. Participants complete paper safety plans as part of their regular treatment, which is a standard of care for suicidal youth.
  Interventions: Behavioral: ASAP (As Safe As Possible); Behavioral: TAU (treatment as usual)
- TAU (treatment as usual) alone (Active Comparator): Participants in this grouping are studied as they proceed from inpatient to outpatient care, per usual treatment protocols at each site. Participants complete paper safety plans as part of their regular treatment, which is a standard of care for suicidal youth.
  Interventions: Behavioral: TAU (treatment as usual)

INTERVENTIONS:
Behavioral: ASAP (As Safe As Possible) — ASAP (As Safe As Possible) is a brief intervention for adolescents hospitalized for suicide risk that focuses on the development of a safety plan, teaching emotion regulation and distress tolerance skills, along with 1-2 post-discharge follow-up calls to encourage adherence to use of the safety plan and to outpatient treatment.
  Arms: ASAP + BRITE + TAU (treatment as usual); ASAP + TAU (treatment as usual)
Behavioral: BRITE smart phone app — BRITE is a smart phone app that aims to support daily emotion regulation and a safety plan that is personalized to the needs and preferences of each adolescent.
  Arms: ASAP + BRITE + TAU (treatment as usual); BRITE + TAU (treatment as usual)
Behavioral: TAU (treatment as usual) — TAU (treatment as usual) is the standard treatment that all adolescents admitted to their respective Inpatient Psychiatry Program receive.

SUMMARY:
In this 2-site study, University of Texas Southwestern Medical Center (UTSW) and Western Psychiatric Institute and Clinic (WPIC), the investigators will conduct a randomized clinical trial (RCT) in 240 psychiatrically hospitalized suicidal adolescents, examining the single and additive effects of two components of an inpatient unit intervention for suicidal adolescents, As Safe As Possible (ASAP), which focuses on emotion regulation and safety planning, and an emotion regulation/safety plan phone app (BRITE).

DETAILED DESCRIPTION:
The investigators aim to randomize 240 adolescents psychiatrically hospitalized for suicidal ideation with a plan or a suicide attempt to one of four treatment arms: (1) ASAP + BRITE + TAU (treatment as usual); (2) BRITE + TAU (treatment as usual); (3) ASAP + TAU (treatment as usual); and (4) TAU (treatment as usual) alone. The investigators will assess suicidal ideation and behavior at 4, 12, and 24 weeks post-intake, in order to:

1. Assess the relative efficacy of ASAP, BRITE and the combination on suicidal ideation, non-suicidal self-injury (NSSI), and suicide attempts, and re-hospitalizations.
2. Examine mediators and moderators of treatment outcome.
3. Examine the costs and cost efficacy of ASAP and BRITE and the combination.

ELIGIBILITY:
Inclusion Criteria:

* Youth admitted to the inpatient unit at either site for a recent suicide attempt or significant suicidal ideation with a plan or intent.
* The youth and parent are able to complete assessments in English, and the youth is able to complete therapy.

Exclusion Criteria:

* The youth currently exhibits psychosis.
* The youth currently exhibits mania.
* The youth is currently <85% of their ideal body weight.
* The youth is intellectually incapable of completing the study, e.g. has an intelligence quotient (IQ) < 70.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 241 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth D. Kennard, PsyD, Principal Investigator — University of Texas Southwestern Medical Center; David A Brent, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kennard BD, Goldstein T, Foxwell AA, McMakin DL, Wolfe K, Biernesser C, Moorehead A, Douaihy A, Zullo L, Wentroble E, Owen V, Zelazny J, Iyengar S, Porta G, Brent D. As Safe as Possible (ASAP): A Brief App-Supported Inpatient Intervention to Prevent Postdischarge Suicidal Behavior in Hospitalized, Suicidal Adolescents. Am J Psychiatry. 2018 Sep 1;175(9):864-872. doi: 10.1176/appi.ajp.2018.17101151. Epub 2018 Jul 19. PMID 30021457
- [Background] Kennard BD, Biernesser C, Wolfe KL, Foxwell AA, Craddock Lee SJ, Rial KV, Patel S, Cheng C, Goldstein T, McMakin D, Blastos B, Douaihy A, Zelazny J, Brent DA. Developing a Brief Suicide Prevention Intervention and Mobile Phone Application: a Qualitative Report. J Technol Hum Serv. 2015 Oct 1;33(4):345-357. doi: 10.1080/15228835.2015.1106384. Epub 2015 Dec 14. PMID 26977137
- [Derived] Goldstein TR, Kennard BD, Porta G, Miller AO, Aguilar K, Bigley K, Vaughn-Coaxum RA, McMakin DL, Douaihy A, Iyengar S, Biernesser CL, Zelazny J, Brent DA. Bridging Gaps in Care Following Hospitalization for Suicidal Adolescents: As Safe As Possible (ASAP) and BRITE App. J Am Acad Child Adolesc Psychiatry. 2025 May;64(5):612-624. doi: 10.1016/j.jaac.2024.06.008. Epub 2024 Jul 18. PMID 39032815

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 241 adolescents were randomized. One randomization accidentally occurred before completion of the baseline assessment, and the participant withdrew consent prior to starting the intervention. No data were collected for this participant. Thus, this report includes 240 adolescents.
Period: Overall Study
Arm/Group | ASAP + BRITE + TAU (Treatment as Usual) | BRITE + TAU (Treatment as Usual) | ASAP + TAU (Treatment as Usual) | TAU (Treatment as Usual) Alone
Started | 60 | 58 | 61 | 61
Completed | 53 | 56 | 55 | 57
Not Completed | 7 | 2 | 6 | 4

BASELINE CHARACTERISTICS:
Population: A total of 241 adolescents were randomized. One randomization accidentally occurred before completion of the baseline assessment, and the participant withdrew consent prior to starting the intervention. No data were collected for this participant. Thus, this report includes 240 adolescents.
Groups:
- Total: Total of all reporting groups
Arm/Group | ASAP + BRITE + TAU (Treatment as Usual) | BRITE + TAU (Treatment as Usual) | ASAP + TAU (Treatment as Usual) | TAU (Treatment as Usual) Alone | Total
Number analyzed (Participants) | 60 | 58 | 61 | 61 | 240
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 60 | 58 | 61 | 61 | 240
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.67 (1.5) | 14.74 (1.57) | 14.52 (1.57) | 14.57 (1.59) | 14.62 (1.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 47 | 53 | 47 | 194
  Male | 13 | 11 | 8 | 14 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 14 | 11 | 9 | 48
  Not Hispanic or Latino | 45 | 43 | 50 | 51 | 189
  Unknown or Not Reported | 1 | 1 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 1 | 2 | 0 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 7 | 6 | 9 | 28
  White | 42 | 42 | 47 | 46 | 177
  More than one race | 7 | 3 | 3 | 3 | 16
  Unknown or Not Reported | 4 | 4 | 4 | 2 | 14
Region of Enrollment [Number; unit: participants]
  United States | 60 | 58 | 61 | 61 | 240
Number of Participants with Actual Suicide Attempts and Suicide Events in Past 3 Months [Count of Participants; unit: Participants] — Actual Attempts: Measured by the CSSRS = Columbia-Suicide Severity Rating Scale
  Suicide Events: Suicidal events were operationalized as any suicide attempt (actual, interrupted, and/or aborted) and/or re-hospitalization over follow-up.Re-hospitalization was assessed at follow-up using the Child and Adolescent Services Assessment (CASA), 37 defined as any inpatient hospitalization in a psychiatric hospital, a psychiatric unit in a general hospital, or a medical inpatient unit for emotional, behavioral, or substance use problems.
  Participants
    Actual attempts in past 3 months | 45 | 38 | 37 | 39 | 159
    Suicide events in past 3 months | 53 | 48 | 46 | 47 | 194

OUTCOME MEASURES:

1. Primary Outcome: Participants With Actual Suicide Attempts as Defined by Columbia Suicide Severity Rating Scale (C-SSRS)
Description: Compare the 4 cells on the rate of actual suicide attempts and time to suicide attempt. Suicide attempt assessed with the Columbia Suicide Severity Rating Scale (C-SSRS)
Time Frame: 1 - 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | ASAP + BRITE + TAU (Treatment as Usual) | BRITE + TAU (Treatment as Usual) | ASAP + TAU (Treatment as Usual) | TAU (Treatment as Usual) Alone
Number analyzed (Participants) | 53 | 56 | 55 | 57
Participants | 6 | 11 | 12 | 10
Statistical Analysis 1: Comparison: ASAP + BRITE + TAU (Treatment as Usual) vs BRITE + TAU (Treatment as Usual) vs ASAP + TAU (Treatment as Usual) vs TAU (Treatment as Usual) Alone; Compare participants receiving ASAP (ASAP+TAU and ASAP+BRITE+TAU) to those who do not (BRITE+TAU and TAU) on the rate of actual suicide attempts; Test type: Superiority; p = 0.71, Chi-squared — False Discovery Rate q-value > 0.99
Statistical Analysis 2: Comparison: ASAP + BRITE + TAU (Treatment as Usual) vs BRITE + TAU (Treatment as Usual) vs ASAP + TAU (Treatment as Usual) vs TAU (Treatment as Usual) Alone; Compare participants receiving BRITE (BRITE+TAU and ASAP+BRITE+TAU) to those who do not (ASAP+TAU and TAU) on the rate of actual suicide attempts; Test type: Superiority; p = 0.43, Chi-squared — False Discovery Rate q-vale > 0.99
Statistical Analysis 3: Comparison: ASAP + BRITE + TAU (Treatment as Usual) vs BRITE + TAU (Treatment as Usual) vs ASAP + TAU (Treatment as Usual) vs TAU (Treatment as Usual) Alone; Compare the 4 arms on the rate of actual suicide attempts in a 2x2 factorial design. Interaction effect of ASAP and BRITE; Test type: Superiority; p = 0.21, Regression, Logistic — False Discovery Rate q-value > 0.99; Odds Ratio (OR) = 0.40, 95% CI 2-sided [0.10 to 1.66]
Statistical Analysis 4: Comparison: ASAP + BRITE + TAU (Treatment as Usual) vs BRITE + TAU (Treatment as Usual) vs ASAP + TAU (Treatment as Usual) vs TAU (Treatment as Usual) Alone; Compare the 4 arms on the rate of actual suicide attempts in a 2x2 factorial design. Main effect of ASAP; Test type: Superiority; p = 0.57, Regression, Logistic — False Discovery Rate q-value > 0.99; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.51 to 3.34]
Statistical Analysis 5: Comparison: ASAP + BRITE + TAU (Treatment as Usual) vs BRITE + TAU (Treatment as Usual) vs ASAP + TAU (Treatment as Usual) vs TAU (Treatment as Usual) Alone; Compare the 4 arms on the rate of actual suicide attempts in a 2x2 factorial design. Main effect of BRITE; Test type: Superiority; p = 0.77, Regression, Logistic — False Discovery Rate q-value > 0.99; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.44 to 2.97]
Statistical Analysis 6: Comparison: ASAP + BRITE + TAU (Treatment as Usual) vs BRITE + TAU (Treatment as Usual) vs ASAP + TAU (Treatment as Usual) vs TAU (Treatment as Usual) Alone; Compare participants receiving ASAP (ASAP+TAU and ASAP+BRITE+TAU) to those who do not (BRITE+TAU and TAU) on time to actual suicide attempt; Test type: Superiority; p = 0.74, Regression, Cox — False Discovery Rate q-value > 0.99; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.48 to 1.69]
Statistical Analysis 7: Comparison: ASAP + BRITE + TAU (Treatment as Usual) vs BRITE + TAU (Treatment as Usual) vs ASAP + TAU (Treatment as Usual) vs TAU (Treatment as Usual) Alone; Compare participants receiving BRITE (BRITE+TAU and ASAP+BRITE+TAU) to those who do not (ASAP+TAU and TAU) on the time to actual suicide attempt; Test type: Superiority; p = 0.45, Regression, Cox — False Discovery Rate q-vale > 0.99; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.42 to 1.48]
Statistical Analysis 8: Comparison: ASAP + BRITE + TAU (Treatment as Usual) vs BRITE + TAU (Treatment as Usual) vs ASAP + TAU (Treatment as Usual) vs TAU (Treatment as Usual) Alone; Compare the 4 arms on time to actual suicide attempt in a 2x2 factorial design. Interaction effect of ASAP and BRITE; Test type: Superiority; p = 0.25, Regression, Cox — False Discovery Rate q-value > 0.99; Hazard Ratio (HR) = 0.47, 95% CI 2-sided [0.13 to 1.72]
Statistical Analysis 9: Comparison: ASAP + BRITE + TAU (Treatment as Usual) vs BRITE + TAU (Treatment as Usual) vs ASAP + TAU (Treatment as Usual) vs TAU (Treatment as Usual) Alone; Compare the 4 arms on time to actual suicide attempt in a 2x2 factorial design. Main effect of ASAP; Test type: Superiority; p = 0.62, Regression, Cox — False Discovery Rate q-value > 0.99; Hazard Ratio (HR) = 1.24, 95% CI 2-sided [0.54 to 2.87]
Statistical Analysis 10: Comparison: ASAP + BRITE + TAU (Treatment as Usual) vs BRITE + TAU (Treatment as Usual) vs ASAP + TAU (Treatment as Usual) vs TAU (Treatment as Usual) Alone; Compare the 4 arms on time to actual suicide attempt in a 2x2 factorial design. Main effect of BRITE; Test type: Superiority; p = 0.83, Regression, Cox — False Discovery Rate q-value > 0.99; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.47 to 2.59]

2. Primary Outcome: Suicidal Events
Description: Defined as actual, aborted, or interrupted attempt based on the the Columbia-Suicide Severity Rating Scale (C-SSRS), and or rehospitalization.
Time Frame: 1 to 24 weeks
Measure: Number; unit: events
Arm/Group | ASAP + BRITE + TAU (Treatment as Usual) | BRITE + TAU (Treatment as Usual) | ASAP + TAU (Treatment as Usual) | TAU (Treatment as Usual) Alone
Number analyzed (Participants) | 54 | 55 | 55 | 57
events | 12 | 23 | 18 | 17
Statistical Analysis 1: Comparison: ASAP + BRITE + TAU (Treatment as Usual) vs BRITE + TAU (Treatment as Usual) vs ASAP + TAU (Treatment as Usual) vs TAU (Treatment as Usual) Alone; Compare participants receiving ASAP (ASAP+TAU and ASAP+BRITE+TAU) to those who do not (BRITE+TAU and TAU) on the rate of suicidal events; Test type: Superiority; p = 0.19, Chi-squared — False Discovery Rate q-value = 0.72; We used standard univariate statistics to compare partici- pants' baseline sociodemographics and clinical characteris- tics by arm [(ASAP vs No ASAP where comparison is 6 www.jaacap.org (ASAP+TAU) and (ASAP+BRITE+TAU) vs (TAU alone) and (BRITE+TAU); and BRITE vs No BRITE where comparison is (ASAP+BRITE+TAU) and (BRITE+TAU) vs (ASAP+TAU) and (TAU Alone)], site, retention, pre- post-COVID and recruitment venue. We then tested for equality of the 2 cells (ASAP vs no ASAP, BRITE vs no BRITE) or 4 cells (ASAP+BRITE+TAU vs BRITE +TAU vs ASAP+TAU vs TAU Alone) without covariates on the rates of and time to suicidal behavior using the appropriate (t or F, c2, Kaplan-Meier, Cox models) test statistics. We then used mixed-effects regression models with arm (2 and 4 cells), time, and their interaction for continuous data. Presented percentages are based on all observed data
Statistical Analysis 2: Comparison: ASAP + BRITE + TAU (Treatment as Usual) vs BRITE + TAU (Treatment as Usual) vs ASAP + TAU (Treatment as Usual) vs TAU (Treatment as Usual) Alone; Compare participants receiving BRITE (BRITE+TAU and ASAP+BRITE+TAU) to those who do not (ASAP+TAU and TAU) on the rate of suicidal events; Test type: Superiority; p = 0.89, Chi-squared — False Discovery Rate q-value > 0.99
Statistical Analysis 3: Comparison: ASAP + BRITE + TAU (Treatment as Usual) vs BRITE + TAU (Treatment as Usual) vs ASAP + TAU (Treatment as Usual) vs TAU (Treatment as Usual) Alone; Compare participants the 4 arms on the rate of suicidal events in a 2x2 factorial design. Interaction effect of ASAP and BRITE; Test type: Superiority; p = 0.08, Regression, Logistic — False Discovery Rate q-value = 0.72; Odds Ratio (OR) = 0.35, 95% CI 2-sided [0.11 to 1.10]
Statistical Analysis 4: Comparison: ASAP + BRITE + TAU (Treatment as Usual) vs BRITE + TAU (Treatment as Usual) vs ASAP + TAU (Treatment as Usual) vs TAU (Treatment as Usual) Alone; Compare the 4 arms on time to actual suicide attempt in a 2x2 factorial design. Main effect of ASAP; Test type: Superiority; p = 0.74, Regression, Logistic — False Discovery Rate q > 0.99; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.51 to 2.55]
Statistical Analysis 5: Comparison: ASAP + BRITE + TAU (Treatment as Usual) vs BRITE + TAU (Treatment as Usual) vs ASAP + TAU (Treatment as Usual) vs TAU (Treatment as Usual) Alone; Compare the 4 arms on time to actual suicide attempt in a 2x2 factorial design. Main effect of BRITE; Test type: Superiority; p = 0.19, Regression, Logistic — False Discovery Rate q=0.72; Odds Ratio (OR) = 1.69, 95% CI 2-sided [0.77 to 3.69]

ADVERSE EVENTS:
Time Frame: up to 24 weeks
Arm/Group | ASAP + BRITE + TAU (Treatment as Usual) | BRITE + TAU (Treatment as Usual) | ASAP + TAU (Treatment as Usual) | TAU (Treatment as Usual) Alone
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/58 | 0/61 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/58 | 0/61 | 1/61
Other Adverse Events (participants affected / at risk) | 0/60 | 0/58 | 1/61 | 1/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASAP + BRITE + TAU (Treatment as Usual) (N=60) | BRITE + TAU (Treatment as Usual) (N=58) | ASAP + TAU (Treatment as Usual) (N=61) | TAU (Treatment as Usual) Alone (N=61)
Suicide Attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Suicide attempt and hospitalized for broken neck
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASAP + BRITE + TAU (Treatment as Usual) (N=60) | BRITE + TAU (Treatment as Usual) (N=58) | ASAP + TAU (Treatment as Usual) (N=61) | TAU (Treatment as Usual) Alone (N=61)
Emergency Room Visit (Social circumstances) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Sexual assault

LIMITATIONS AND CAVEATS:
Methods were modified with treatment delivered virtually post hospital discharge due to COVID. Limited diversity of the sample may reflect substantial disparities in mental health service provision for suicidal youth.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/88/NCT03825588/Prot_SAP_000.pdf